CLINICAL TRIAL: NCT00770029
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Investigate the Efficacy and Safety of IncobotulinumtoxinA (Xeomin), Free of Complexing Proteins, in the Treatment of Glabellar Frown Lines. No. 2
Brief Title: IncobotulinumtoxinA (Xeomin) Versus Placebo in the Treatment of Glabellar Frown Lines No. 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201 - 0724 / 1
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Moderate to Severe Glabellar Frown Lines
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IncobotulinumtoxinA (Xeomin) (20 Units) (Experimental): IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150 kD), free from complexing proteins' (active ingredient: Clostridium Botulinum neurotoxin type A free from complexing proteins) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% sodium chloride (NaCl), 20 units, total volume 0.5 mL, mode of administration: intramuscular injection
  Interventions: Drug: IncobotulinumtoxinA (Xeomin) (20 Units)
- Placebo (Placebo Comparator): Placebo to IncobotulinumtoxinA (Xeomin) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl, corresponding to total placebo volume 0.5 mL; mode of administration: intramuscular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IncobotulinumtoxinA (Xeomin) (20 Units) — The treatment will be administered only once at day 0 at five injection sites in the glabellar area. The total dose of 20 Units IncobotulinumtoxinA (Xeomin) is reconstituted in a total injection volume of 0.5 mL that is to be injected to the five sites in equal aliquots of 0.1 mL.
  Other Names: IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150 kD), free from complexing proteins' (20 Units)
  Arms: IncobotulinumtoxinA (Xeomin) (20 Units)
Drug: Placebo — The treatment will be administered only once at day 0 at five injection sites in the glabellar area. Volume of Placebo equivalent to IncobotulinumtoxinA (Xeomin).
  Arms: Placebo

SUMMARY:
The study objective was to show the superior efficacy of IncobotulinumtoxinA (Xeomin) over placebo by evaluation of treatment success analyzing the investigator's rating on the Facial Wrinkle Scale and the patient's assessment on a 4-point scale. 255 female and male patients with moderate to severe glabellar frown lines to be randomized in a 2:1 ratio to receive one injection of IncobotulinumtoxinA (Xeomin) or placebo and will be followed up until day 120.

DETAILED DESCRIPTION:
The study was a prospective, randomized, double-blind, placebo-controlled, parallel-group, multicenter phase 3 clinical trial. Approximately 285 females and males with moderate to severe glabellar frown lines at maximum frown were to be screened during a screening period of four months in order to randomize approximately 255 subjects into one treatment and one placebo group at a ratio of 2 : 1. After the single injection treatment with a total dose of 20 Units IncobotulinumtoxinA (Xeomin) or corresponding placebo, the subjects were observed over 120 days. During the study participation the subjects performed seven visits.

Eight (8) sites in the United States and Canada participated in this trial. The study was led by one Lead PI and a Co-Lead PI who was assisting the Lead PI. The role of the Lead PI and the Co-Lead PI was executed by one of the PIs of this study, respectively. The PI at each site was a medical doctor who was experienced in aesthetic dermatology, i.e. who had several years (>=2 years) of experience in treatment of glabellar frown lines with BTX-A preparations. The PI was the person who led the team at one trial site and who was responsible for the conduct of the clinical trial at the site. The sub-investigator was a member of the team designated by the PI to perform important trial-related decisions. A maximum number of two sub-investigators could be authorized for injection and rating if necessary. At each site, ideally one investigator was to inject and rate all subjects. Injecting and rating sub-investigators had to be medical doctors with several years of experience in treatment of glabellar frown lines with BTX-A preparations. A subject had to be rated by the same investigator at all visits. Another phase 3 trial MRZ 60201-0741/1 (NCT00770211) with design and endpoints identical to those in this trial was performed in order to compare efficacy and safety results with a second study population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Moderate to severe glabellar frown lines at maximum frown (severity score of 2 or 3 on Facial Wrinkle Scale as assessed by investigator's rating: 0= 'none', 1= 'mild', 2= 'moderate', 3= 'severe'
* Moderate to severe glabellar frown lines at maximum frown (severity score of 2 or 3 on Facial Wrinkle Scale as assessed by patient's assessment: 0= 'none', 1= 'mild', 2= 'moderate', 3= 'severe'
* Stable medical condition

Exclusion Criteria:

* Previous treatment with Botulinum toxin of any serotype in the glabellar area within the last 8 month
* Previous treatment with any facial aesthetic procedure (e.g. injection with biodegradable fillers, chemical peeling, photo rejuvenation) in the glabellar area within the last 12 month
* Previous insertion of permanent material in the glabellar area (regardless of the time between previous treatment and this study)
* Planned treatment with Botulinum toxin of any serotype in any other body region during the study period
* Any surgery in the glabellar area including surgical removal of the corrugator, procerus, or depressor supercilii muscles or a combination of these, or scars in the glabellar area and the surrounding areas (including eye brow)
* Any other planned facial aesthetic procedure during the trial period
* Inability to substantially lessen glabellar frown lines even by physically spreading them apart
* Marked facial asymmetry or ptosis of eyelid and/or eyebrow
* History of facial nerve palsy
* Any infection in the area of the injection sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Carruthers, MD, Principal Investigator; Jean Carruthers, MD, Principal Investigator
Locations (8):
- United States (5):
  - Skin Care Center, Los Angeles, California
  - Coleman William, Meatrie, Louisiana
  - SkinCare Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - Flynn Consulting PLLC, Raleigh, North Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
- Canada (3):
  - Aesthetic Facial Ophtalmology, Vancouver, British Columbia
  - Carruthers Clinical Research, Vancouver, British Columbia
  - Solish Nowell, Toronto, Ontario

REFERENCES:
- [Result] Carruthers A, Carruthers J, Coleman WP 3rd, Donofrio L, Flynn T, Gold M, Heinz M, Harrington L, Jones D, McDaniel D, Rohrer T, Schlobe A, Solish N, Weiss RA. Multicenter, randomized, phase III study of a single dose of incobotulinumtoxinA, free from complexing proteins, in the treatment of glabellar frown lines. Dermatol Surg. 2013 Apr;39(4):551-8. doi: 10.1111/dsu.12100. Epub 2013 Feb 4. PMID 23379292

RESULTS

PARTICIPANT FLOW:
Groups:
- IncobotulinumtoxinA (Xeomin) (20 Units): IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150 kD), free from complexing proteins' (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection, 20 units; mode of administration: intramuscular injection
- Placebo: Placebo to IncobotulinumtoxinA (Xeomin) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl; mode of administration: same as for IncobotulinumtoxinA (Xeomin).
Period: Overall Study
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo
Started | 184 | 92
Completed | 178 | 89
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo | Total
Number analyzed (Participants) | 184 | 92 | 276
Age Continuous [Mean (Standard Deviation); unit: years] | 46.6 (9.87) | 46.4 (10.56) | 46.6 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 76 | 238
  Male | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint Treatment Success (CETS) Constituted by 2 Variables: 2-point Responders at Maximum Frown (Frown as Much as Possible) at Day 30 by Investigator's Rating on Facial Wrinkle Scale (FWS) and by Patient's Assessment on 4-point Scale
Description: Composite endpoint CETS constituted by two efficacy variables:
  1. The investigator's assessment on the four-point FWS: none = 0, mild = 1, moderate = 2, severe = 3.
  2. Patient's assessment on the 4-point scale in comparison to sample photos: 0 = No muscle action at all; 1 = Some even slight muscle action possible i.e. visible furrows; 2 = Moderately strong muscle action possible i.e. visible muscle bulges; 3 = Strong muscle action possible which may cause local pallor.
  A subject was a responder only if a 2-point improvement compared to baseline occurred simultaneously for both variables.
Time Frame: Baseline to Day 30
Population: Full Analysis Set (FAS): All randomized subjects treated with study medication. Missing values were imputed by the evaluations made at Day 7 according to the LOCF (last observation carried forward). If no ratings for Day 7 were available values were set to 'no 2-point responder'.
Measure: Number; unit: Participants
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo
Number analyzed (Participants) | 184 | 92
Participants | 111 | 0
Statistical Analysis 1: Comparison: IncobotulinumtoxinA (Xeomin) (20 Units) vs Placebo; The efficacy of the treatment was confirmed if H0 was rejected at a given α of 5%, that means if the two sided p-value was ≤0.05. Power of 90%; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Difference response rate = 0.60, 95% CI 2-sided [0.52 to 0.68], Standard Error of Mean 0.036

2. Secondary Outcome: Responders at Rest at Day 30 by Investigator's Rating on FWS.
Description: The investigator's assessment at rest (no muscle action in the face, no frown at all) on the four-point FWS: none = 0, mild = 1, moderate = 2, severe = 3. A responder was defined as a subject with a rating of none = 0 or mild = 1.
Time Frame: Baseline to Day 30
Population: The number and percentage of responses by treatment group will be provided for all secondary endpoints on the FAS observed cases.
Measure: Number; unit: Participants
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo
Number analyzed (Participants) | 184 | 92
Participants | 123 | 36

3. Secondary Outcome: 1-point Responders at Rest at Day 30 by Patient's Assessment on 4-point Scale.
Description: Patient's assessment at rest (no muscle action in the face, no frown at all) on the 4-point scale in comparison to sample photos: 0 = No visible vertical line(s) at all (i.e. no visible upright line); 1 = Slightly visible vertical line(s) (i.e. slightly visible upright line); 2 = Moderate vertical line(s) with depression (i.e. upright line with deepening); 3 = Deep vertical line(s) and depression which cannot be effaced by spreading (i.e. cannot be smoothed out).
  A subject was a responder if a 1-point improvement occurred compared to baseline.
Time Frame: Baseline to Day 30
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo
Number analyzed (Participants) | 184 | 92
Participants | 131 | 10

4. Secondary Outcome: Responders at Maximum Frown at Day 30 by Investigator's Rating on FWS.
Description: The investigator's assessment at maximum frown (frown as much as possible) on the four-point FWS: none = 0, mild = 1, moderate = 2, severe = 3. A responder was defined as a subject with a rating of none = 0 or mild = 1.
Time Frame: Baseline to Day 30
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo
Number analyzed (Participants) | 184 | 92
Participants | 147 | 0

5. Secondary Outcome: 1-point Responders at Maximum Frown at Day 30 by Patient's Assessment on 4-point Scale.
Description: Patient's assessment at maximum frown (frown as much as possible) on the 4-point scale in comparison to sample photos: 0 = No muscle action at all; 1 = Some even slight muscle action possible i.e. visible furrows; 2 = Moderately strong muscle action possible i.e. visible muscle bulges; 3 = Strong muscle action possible which may cause local pallor.
  A subject was a responder if a 1-point improvement occurred compared to baseline.
Time Frame: Baseline to Day 30
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo
Number analyzed (Participants) | 184 | 92
Participants | 161 | 9

ADVERSE EVENTS:
Time Frame: All SAEs/AEs after injection were reported. All subjects experiencing SAEs/AEs were to be monitored until AE was resolved or stabilized or until a plausible explanation for the cause of the event had been found.
Description: Data pertaining to AEs were collected during each study visit either based on the subject's spontaneous description or by investigator's inquiry or discovered in the course of examinations done during the visit. The table of 'Other Adverse Events' includes all non-serious AEs.
Arm/Group | IncobotulinumtoxinA (Xeomin) (20 Units) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/184 | 1/92
Other Adverse Events (participants affected / at risk) | 32/184 | 15/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IncobotulinumtoxinA (Xeomin) (20 Units) (N=184) | Placebo (N=92)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Start date: 23JAN2009 Stop date: 21JUL2009 Mild in intensity Not related to study treatment Recovered/resolved
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Start date: 23JAN2009 Stop date: 21JUL2009 Mild in intensity Not related to study treatment Recovered/resolved
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — AE leading to withdrawal
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IncobotulinumtoxinA (Xeomin) (20 Units) (N=184) | Placebo (N=92)
Nasopharyngitis (Infections and infestations) | 10 (10) | 5 (5)
Headache (Nervous system disorders) | 13 (13) | 6 (7)
Sinusitis (Infections and infestations) | 6 (6) | 3 (3)
Bronchitis (Infections and infestations) | 4 (5) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results to be published without written agreement by sponsor; manuscripts to be sent to sponsor at least 6 wks before submission. Sponsor to give written opinion within 30 d. Sponsor is entitled to exert influence on the contents of publications, to postpone publications up to 36 months after end of the study, and to name co-authors. In case of justified doubts of sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.